CLINICAL TRIAL: NCT05661292
Title: Validation of Advanced Colorectal Neoplasm Risk Categories in Screening Colonoscopy and Identification of Biomarkers in a Prospective Cohort in Mexico.
Brief Title: Validation of Advanced Colorectal Neoplasm Risk Categories in a Prospective Cohort in Mexico
Acronym: COLOFIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, David Huitzil m, Medical Doctor, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: HEM-2756-18-21-1
Record Dates: First submitted 2022-03-04; First posted 2022-12-22 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal cancer; Screening; Mexico
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Blood Specimen Collection; Urination; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This is an optional research. If the subject accept to participate, we will get and store:
  1. Blood: 15 ml
  2. Urine: 20 ml
  3. Tissue samples: just when biopsies were taken in the colonoscopy for diagnostic purposes. No additional biopsies not required for medical attention will be taken. These tissue samples will be used just when they are not required to stablish a diagnosis.
  All these samples will be storage and used for future biomedical research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fecal inmunochemical test — A fecal inmunochemical test will be performed prior to colonoscopy.
  Other Names: FIT
Diagnostic Test: Colonoscopy — A colonoscopy will be performed. Any polyp identified will be resected (polypectomy) and analyzed histologically. NOTE: The subject and colonoscopist will be blinded to FIT test results and risk category.
Biological: Optional collection of tissue, blood and urine for future biomedical research — Subjects may optionally participate in the collection of tissue, blood, and urine samples for future biomedical research. This procedure consists of taking a 15 ml sample of venous blood and 20 ml of urine. The tissue samples to be used will be those that have been taken for diagnostic purposes during the colonoscopy. Additional biopsies not required for medical care will not be taken. These samples will be used as long as they are no longer required to establish a diagnosis.
  Other Names: Tissue, blood and urine

SUMMARY:
Worldwide, there are 1,361,000 new cases of colorectal cancers (CRC) annually, with 694,000 deaths. However, the incidence varies by up to a factor of 10x between high and low incidence countries (eg. USA vs Mexico, incidence rate of 42.54 vs 7.44 / 100,000 inhabitants). Mexico is considered a low-incidence country, with 8,651 new cases and 4,694 deaths annually.

CRC is a preventable and detectable disease. Screening programs established in high-incidence countries have managed to reduce the incidence and mortality from this disease and it is considered a cost-effective strategy. In less developed countries where there are no screening programs for CRC, the highest number of deaths occurs despite having the lowest number of cases. It is recognized that a barrier to establishing a screening program in a country with low incidence and limited resources is cost-effectiveness.

The prevalence of Advanced Colorectal Neoplasia (ACN) detected by screening colonoscopy in a Mexican cohort of 1172 INNSZ patients was 2.9%. In the US the prevalence is 7.6%. The number of colonoscopies to be performed to detect ACN was estimated at 34 for Mexico and 13 for the US, which suggests that the cost-effectiveness of screening colonoscopy could be 3 times lower in our country.

In Mexico there is no national screening program for CRC. The eligible population (adults between 50 and 75 years old) for CRC screening is estimated in 20 million of Mexicans. It is recognized that Mexico does not have enough financial resources nor the infrastructure to screen the entire eligible population either by direct colonoscopy, or by FIT (fecal immunochemical test) followed by colonoscopy. With a 5% frequency of positive FIT, nearly 1,000,000 follow-up colonoscopies would be required annually in a population screening program.

An alternative could be to offer screening based on risk, which means only offering screening to the highest-risk population.

There are calculators to predict the risk of identifying ACN in a screening colonoscopy, however, none have been developed and validated in the Mexican population. The weight of the risk factors associated with ACN in the Mexican population could be different, so it is necessary to develop and validate an ACN risk calculator that allows the Mexican population to be stratified and to concentrate screening efforts on the population at highest risk.

DETAILED DESCRIPTION:
This is a prospective cohort of subjects eligible for CRC screening in Mexico City.

The main goal is to validate the APCS clinical score as a risk - stratification tool for screening colonoscopy in a Mexican population.

The Asian-Pacific Colorectal Screening (APCS) score is a clinical tool used to stratify subjects according to the probability of identification of Advanced Colorectal Neoplasia (ACN) in a screening colonoscopy. ACN includes lesions larger than 10 mm with one or more of the following: a villous content, high-grade dysplasia, or carcinoma. The tool stratifies the population into three risk categories, considering: age, sex, smoking history, and first-degree family history of colorectal cancer. The total score obtained allows the stratification into average risk (0-1 point), moderate (2-3 points), and high risk (4-7 points). The prevalence of ACN in the original validation cohort of the APCS was 1.3% for average risk, 3.2% in moderate risk and 5.2% in high risk.

Investigators previously evaluated the APCS score in a retrospective study of screening colonoscopy in Mexican population (n=1269). The prevalence of ACN was 2.6% vs 5.2% (p=0.027) for moderate risk and high-risk categories, respectively.

To implement a risk-stratified screening program for the Mexican population, prospective validation was considered necessary. A prospective study would allow for collection and evaluation of additional variables that could potentially improve APCS score. FIT cut-off values have never been validated in Mexican population and are required to implement a national colorectal screening program. Prospective design will also allow for bio banking for future medical research.

The following procedures will be performed:

1. Subjects will be invited to participate in the study, and if they accept, an informed consent will be given and explained to them. They will have a standardized interview dedicated to promoting CRC screening and complete a CRC risk factor questionnaire to determine their risk category.
2. Subjects may optionally participate in the collection of tissue, blood, and urine samples for future biomedical research. This procedure consists of taking a 15 ml sample of venous blood and 20 ml of urine. The tissue samples to be used will be those that have been taken for diagnostic purposes during the colonoscopy. Additional biopsies not required for medical care will not be taken. These samples will be used as long as they are no longer required to establish a diagnosis.
3. A Fecal Immunochemical Test (FIT) will be performed prior to the colonoscopy. Note: A positive FIT will have a Hb value >20 ug/g of stool.
4. A colonoscopy will be performed. Any polyp identified will be resected (polypectomy) and analyzed histologically. NOTE: The subject and physician will be blinded to FIT test results and risk category.

   In subsequent medical consultation, the results of the risk score, the FIT test, and colonoscopy will be discussed.
5. If the patient does not perform any of the tests, they will be interviewed on a second occasion to complete a questionnaire of reasons of rejection. NOTE: It is anticipated that a proportion of subjects will verbally accept the screening, but the proposed tests will not be carried out (this will measure the percentage of acceptance of the recommendation).

Given that age and gender are the most important risk factors, the population will be stratified simulating the Mexican population pyramid as follows: 50% male subjects and 50% female subjects. By age groups: 50-54 years (31%), 55-59 (24%), 60-64 (19%), 65-69 (14%), 70-75 (12%).

The data collected from the participants will be entered into an electronic registry (Redcap) in real-time. A periodic review of the electronic registry will be carried out by personal of the protocol to ensure the quality of the information and that it is complete. The study does not contemplate external monitoring of the data.

Statistical considerations

* Sample size: for a difference in proportions of 2.6% (prevalence of ACN 5.2% vs. 2.6% in the high vs. moderate-risk population), 868 subjects per group are required to achieve a power of 80%, with a confidence level of 95 %, that is, 1736 subjects. It is anticipated that in 15% of the subjects the two screening tests will not be available, so a total sample of 2000 subjects is proposed.
* Statistical proportions, means, and medians will be used to describe the population. The differences in proportions will be analyzed with the X2 test. Using a binary logistic regression model, variables associated with ACN risk will be identified. A p < 0.05 will be considered statistically significant. The risk calculator will be developed using the variables identified in the univariate analysis and differential weight will be assigned to them according to risk. To determine the optimal cut-off point in FIT test (ng of hemoglobin per gram of feces): the investigators will use the distribution of the FIT score for patients with and without premalignant lesions and/or colorectal cancer to estimate sensitivity and specificity. according to different cut-off values. Subsequently, the investigators will use a decision model based on specificity/sensitivity ROC curves and according to different FIT cut-off points. The closer the ROC curve is to the upper left corner, the higher the predictive power of detecting colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects between 50 and 75 years of age-eligible for CRC screening with or without registry at the institute.

Note: concerning symptoms of CRC diagnosis will not be admitted: fresh blood in the stool, black stools, unexplained weight loss (>10% of usual body weight). Concerning symptoms of Functional Gastrointestinal Disorder (FGID) will be permitted: loss of appetite, diarrhea, constipation, abdominal pain or discomfort.

* Subjects who give their informed consent.
* Subjects who have completed the vaccination schedule against the SARS CoV-2 virus with any of the vaccines approved in Mexico, at least 4 weeks before the colonoscopy.

Exclusion Criteria:

* Personal history of any type of cancer, except basal cell carcinoma or cervical cancer in situ.
* Personal history of colon polyps.
* Personal history of abdominal or pelvic radiation due to previous cancer.
* Relatives with familial adenomatous polyposis (FAP) or hereditary non-polyposis CRC.
* Inflammatory bowel disease (IBD).
* High anesthetic risk (ASA greater than 3 of the classification of the American Society of Anesthesiology).
* Any medical condition that limits life expectancy at the discretion of the investigator.
* Charlson index > 4.
* Presence of anemia in the last year according to the WHO definition: women <12 g/dl, men <13 g/dl.
* Previous colectomy.
* Colonoscopy in the previous 5 years.
* Sigmoidoscopy in the previous 3 years.
* A fecal occult blood test in the past year.
* CT colonography in the previous 10 years.
* Clinical data suggestive of CRC such as hematochezia, melena, weight loss greater than 10% of usual body weight in a 6 months period.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for CRC screening with or without institutional registry. Subjects with institutional registry will be identified among patients treated at the Internal Medicine clinic of the Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán" in Mexico City. Patients without institutional registry will be identified among relatives of participants, blood bank, and by diffusion of the protocol with leaflets on social networks and internal at our center.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Asian Pacific Colorectal Screening (APCS) score validation in Mexican population. | 3 years
  Estimation of the prevalence of Advanced colorectal neoplasia (ACN) in high-risk category compared to the prevalence of ACN in moderate-risk category according to APCS score in screening colonoscopy. The tool stratifies the population into three risk categories, taking into account: age, sex, smoking history, and first-degree family history of colorectal cancer. The total score obtained allows the stratification into average risk (0-1 point), moderate (2-3 points), and high risk (4-7 points) categories. The prevalence of ACN in the original validation cohort of the APCS was 1.3% for average risk, 3.2% in moderate risk and 5.2% in high risk categories.

SECONDARY OUTCOMES:
Development and validation of a novel risk stratification model to detect Advanced Colorectal Neoplasia (ACN) in Mexican population. | 3 years
  Risk ratio (RR) of variables relevant to Mexican population related to ACN will be identified in prospectively collected clinical questionnaires.
  The variables include:
  demographic data (sex and age), familiar history, presence of diabetes and hypertension, body mass index, smoking history, Non-Steroideal Anti-Inflammatory Drugs (NSAIDs) consumption, diet and physical activity. Selected variables will be incorporated in a new model to have two risk groups, a high and a low risk. Each group defines the risk of find ACN in a screening colonoscopy. The performance of the new model will be evaluated by comparing the RR of ACN in high vs low risk categories.
Optimal Fecal Immunochemical Test (FIT) valued for Advanced Colorectal Neoplasia (ACN) detection. | 3 years
  Hemoglobin per gram of feces to categorize a FIT as positive for ACN detection derived from a Receiver Operating Characteristic (ROC) curve analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel D Huitzil-Melendez, MS, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Not aplicable

REFERENCES:
- [Background] Allison JE, Fraser CG, Halloran SP, Young GP. Population screening for colorectal cancer means getting FIT: the past, present, and future of colorectal cancer screening using the fecal immunochemical test for hemoglobin (FIT). Gut Liver. 2014 Mar;8(2):117-30. doi: 10.5009/gnl.2014.8.2.117. Epub 2014 Mar 11. PMID 24672652
- [Background] Baxter NN, Warren JL, Barrett MJ, Stukel TA, Doria-Rose VP. Association between colonoscopy and colorectal cancer mortality in a US cohort according to site of cancer and colonoscopist specialty. J Clin Oncol. 2012 Jul 20;30(21):2664-9. doi: 10.1200/JCO.2011.40.4772. Epub 2012 Jun 11. PMID 22689809
- [Background] Brenner H, Chang-Claude J, Rickert A, Seiler CM, Hoffmeister M. Risk of colorectal cancer after detection and removal of adenomas at colonoscopy: population-based case-control study. J Clin Oncol. 2012 Aug 20;30(24):2969-76. doi: 10.1200/JCO.2011.41.3377. Epub 2012 Jul 23. PMID 22826281
- [Background] Bujanda L, Cosme A, Gil I, Arenas-Mirave JI. Malignant colorectal polyps. World J Gastroenterol. 2010 Jul 7;16(25):3103-11. doi: 10.3748/wjg.v16.i25.3103. PMID 20593495
- [Background] Chiang TH, Chuang SL, Chen SL, Chiu HM, Yen AM, Chiu SY, Fann JC, Chou CK, Lee YC, Wu MS, Chen HH. Difference in performance of fecal immunochemical tests with the same hemoglobin cutoff concentration in a nationwide colorectal cancer screening program. Gastroenterology. 2014 Dec;147(6):1317-26. doi: 10.1053/j.gastro.2014.08.043. Epub 2014 Sep 6. PMID 25200099
- [Background] Coleman HG, Loughrey MB, Murray LJ, Johnston BT, Gavin AT, Shrubsole MJ, Bhat SK, Allen PB, McConnell V, Cantwell MM. Colorectal Cancer Risk Following Adenoma Removal: A Large Prospective Population-Based Cohort Study. Cancer Epidemiol Biomarkers Prev. 2015 Sep;24(9):1373-80. doi: 10.1158/1055-9965.EPI-15-0085. Epub 2015 Jun 16. PMID 26082403
- [Background] Eduardo Negrete Carballo, Fidel David Huitzil Melendez. Prevalence of advanced colorectal neoplasia according to risk categories at screening colonoscopy in a tertiary referral center. Journal of Clinical Oncology 36, no. 4_suppl (February 2018) 578-578. DOI: 10.1200/JCO.2018.36.4_suppl.578.
- [Background] Freedman AN, Slattery ML, Ballard-Barbash R, Willis G, Cann BJ, Pee D, Gail MH, Pfeiffer RM. Colorectal cancer risk prediction tool for white men and women without known susceptibility. J Clin Oncol. 2009 Feb 10;27(5):686-93. doi: 10.1200/JCO.2008.17.4797. Epub 2008 Dec 29. PMID 19114701
- [Background] Flitcroft KL, Irwig LM, Carter SM, Salkeld GP, Gillespie JA. Colorectal cancer screening: why immunochemical fecal occult blood tests may be the best option. BMC Gastroenterol. 2012 Dec 29;12:183. doi: 10.1186/1471-230X-12-183. PMID 23272939
- [Background] Fraser CG, Allison JE, Halloran SP, Young GP; Expert Working Group on Fecal Immunochemical Tests for Hemoglobin, Colorectal Cancer Screening Committee, World Endoscopy Organization. A proposal to standardize reporting units for fecal immunochemical tests for hemoglobin. J Natl Cancer Inst. 2012 Jun 6;104(11):810-4. doi: 10.1093/jnci/djs190. Epub 2012 Apr 2. PMID 22472305
- [Background] Guy GP Jr, Richardson LC, Pignone MP, Plescia M. Costs and benefits of an organized fecal immunochemical test-based colorectal cancer screening program in the United States. Cancer. 2014 Aug 1;120(15):2308-15. doi: 10.1002/cncr.28724. Epub 2014 Apr 15. PMID 24737634
- [Background] Hernandez V, Cubiella J, Gonzalez-Mao MC, Iglesias F, Rivera C, Iglesias MB, Cid L, Castro I, de Castro L, Vega P, Hermo JA, Macenlle R, Martinez-Turnes A, Martinez-Ares D, Estevez P, Cid E, Vidal MC, Lopez-Martinez A, Hijona E, Herreros-Villanueva M, Bujanda L, Rodriguez-Prada JI; COLONPREV Study Investigators. Fecal immunochemical test accuracy in average-risk colorectal cancer screening. World J Gastroenterol. 2014 Jan 28;20(4):1038-47. doi: 10.3748/wjg.v20.i4.1038. PMID 24574776
- [Background] Hol L, van Leerdam ME, van Ballegooijen M, van Vuuren AJ, van Dekken H, Reijerink JC, van der Togt AC, Habbema JD, Kuipers EJ. Screening for colorectal cancer: randomised trial comparing guaiac-based and immunochemical faecal occult blood testing and flexible sigmoidoscopy. Gut. 2010 Jan;59(1):62-8. doi: 10.1136/gut.2009.177089. PMID 19671542
- [Background] Hol L, Wilschut JA, van Ballegooijen M, van Vuuren AJ, van der Valk H, Reijerink JC, van der Togt AC, Kuipers EJ, Habbema JD, van Leerdam ME. Screening for colorectal cancer: random comparison of guaiac and immunochemical faecal occult blood testing at different cut-off levels. Br J Cancer. 2009 Apr 7;100(7):1103-10. doi: 10.1038/sj.bjc.6604961. PMID 19337257
- [Background] Howlader N, Noone AM, Krapcho M, et al. SEER Cancer Statistics Review, 1975-2011. Bethesda MD: National Cancer Institute; 2014. http://seer.cancer.gov./csr/1975_2011/, based on November 2013 SEER data submission, posted to the SEER web site.
- [Background] Imperiale TF, Ransohoff DF, Itzkowitz SH, Levin TR, Lavin P, Lidgard GP, Ahlquist DA, Berger BM. Multitarget stool DNA testing for colorectal-cancer screening. N Engl J Med. 2014 Apr 3;370(14):1287-97. doi: 10.1056/NEJMoa1311194. Epub 2014 Mar 19. PMID 24645800
- [Background] Inadomi JM. Screening for Colorectal Neoplasia. N Engl J Med. 2017 Apr 20;376(16):1599-1600. doi: 10.1056/NEJMc1702535. No abstract available. PMID 28423294
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Jenkins PJ, Fairclough PD; British Society for Gastroenterology; Association of Coloproctology for Great Britain and Ireland. Screening guidelines for colorectal cancer and polyps in patients with acromegaly. Gut. 2002 Oct;51 Suppl 5(Suppl 5):V13-4. doi: 10.1136/gut.51.suppl_5.v13. No abstract available. PMID 12221033
- [Background] Langner C. Serrated and non-serrated precursor lesions of colorectal cancer. Dig Dis. 2015;33(1):28-37. doi: 10.1159/000366032. Epub 2014 Dec 17. PMID 25531494
- [Background] Lee JK, Liles EG, Bent S, Levin TR, Corley DA. Accuracy of fecal immunochemical tests for colorectal cancer: systematic review and meta-analysis. Ann Intern Med. 2014 Feb 4;160(3):171. doi: 10.7326/M13-1484. PMID 24658694
- [Background] Levi Z, Rozen P, Hazazi R, Vilkin A, Waked A, Maoz E, Birkenfeld S, Lieberman N, Klang S, Niv Y. Sensitivity, but not specificity, of a quantitative immunochemical fecal occult blood test for neoplasia is slightly increased by the use of low-dose aspirin, NSAIDs, and anticoagulants. Am J Gastroenterol. 2009 Apr;104(4):933-8. doi: 10.1038/ajg.2009.14. Epub 2009 Mar 17. PMID 19293792
- [Background] Muto T, Bussey HJ, Morson BC. The evolution of cancer of the colon and rectum. Cancer. 1975 Dec;36(6):2251-70. doi: 10.1002/cncr.2820360944. PMID 1203876
- [Background] Park DI, Ryu S, Kim YH, Lee SH, Lee CK, Eun CS, Han DS. Comparison of guaiac-based and quantitative immunochemical fecal occult blood testing in a population at average risk undergoing colorectal cancer screening. Am J Gastroenterol. 2010 Sep;105(9):2017-25. doi: 10.1038/ajg.2010.179. Epub 2010 May 25. PMID 20502450
- [Background] Quintero E, Castells A, Bujanda L, Cubiella J, Salas D, Lanas A, Andreu M, Carballo F, Morillas JD, Hernandez C, Jover R, Montalvo I, Arenas J, Laredo E, Hernandez V, Iglesias F, Cid E, Zubizarreta R, Sala T, Ponce M, Andres M, Teruel G, Peris A, Roncales MP, Polo-Tomas M, Bessa X, Ferrer-Armengou O, Grau J, Serradesanferm A, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, de la Vega-Prieto M, Reyes-Melian JM, Cacho G, Diaz-Tasende J, Herreros-de-Tejada A, Poves C, Santander C, Gonzalez-Navarro A; COLONPREV Study Investigators. Colonoscopy versus fecal immunochemical testing in colorectal-cancer screening. N Engl J Med. 2012 Feb 23;366(8):697-706. doi: 10.1056/NEJMoa1108895. PMID 22356323
- [Background] Stegeman I, de Wijkerslooth TR, Stoop EM, van Leerdam M, van Ballegooijen M, Kraaijenhagen RA, Fockens P, Kuipers EJ, Dekker E, Bossuyt PM. Risk factors for false positive and for false negative test results in screening with fecal occult blood testing. Int J Cancer. 2013 Nov 15;133(10):2408-14. doi: 10.1002/ijc.28242. Epub 2013 Jun 25. PMID 23649826
- [Background] van Rossum LG, van Rijn AF, Laheij RJ, van Oijen MG, Fockens P, van Krieken HH, Verbeek AL, Jansen JB, Dekker E. Random comparison of guaiac and immunochemical fecal occult blood tests for colorectal cancer in a screening population. Gastroenterology. 2008 Jul;135(1):82-90. doi: 10.1053/j.gastro.2008.03.040. Epub 2008 Mar 25. PMID 18482589
- [Background] van Turenhout ST, Oort FA, Terhaar sive Droste JS, Coupe VM, van der Hulst RW, Loffeld RJ, Scholten P, Depla AC, Bouman AA, Meijer GA, Mulder CJ, van Rossum LG. Hemorrhoids detected at colonoscopy: an infrequent cause of false-positive fecal immunochemical test results. Gastrointest Endosc. 2012 Jul;76(1):136-43. doi: 10.1016/j.gie.2012.03.169. PMID 22726472
- [Background] Williams JG, Pullan RD, Hill J, Horgan PG, Salmo E, Buchanan GN, Rasheed S, McGee SG, Haboubi N; Association of Coloproctology of Great Britain and Ireland. Management of the malignant colorectal polyp: ACPGBI position statement. Colorectal Dis. 2013 Aug;15 Suppl 2:1-38. doi: 10.1111/codi.12262. No abstract available. PMID 23848492
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Wong MC, Ching JY, Chan VC, Lam TY, Luk AK, Ng SS, Sung JJ. Factors associated with false-positive and false-negative fecal immunochemical test results for colorectal cancer screening. Gastrointest Endosc. 2015 Mar;81(3):596-607. doi: 10.1016/j.gie.2014.08.006. Epub 2014 Oct 5. PMID 25293827
- [Background] Yeoh KG, Ho KY, Chiu HM, Zhu F, Ching JY, Wu DC, Matsuda T, Byeon JS, Lee SK, Goh KL, Sollano J, Rerknimitr R, Leong R, Tsoi K, Lin JT, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. The Asia-Pacific Colorectal Screening score: a validated tool that stratifies risk for colorectal advanced neoplasia in asymptomatic Asian subjects. Gut. 2011 Sep;60(9):1236-41. doi: 10.1136/gut.2010.221168. Epub 2011 Mar 14. PMID 21402615
- [Background] Young GP, Symonds EL, Allison JE, Cole SR, Fraser CG, Halloran SP, Kuipers EJ, Seaman HE. Advances in Fecal Occult Blood Tests: the FIT revolution. Dig Dis Sci. 2015 Mar;60(3):609-22. doi: 10.1007/s10620-014-3445-3. Epub 2014 Dec 10. PMID 25492500
- [Background] Zauber AG. The impact of screening on colorectal cancer mortality and incidence: has it really made a difference? Dig Dis Sci. 2015 Mar;60(3):681-91. doi: 10.1007/s10620-015-3600-5. Epub 2015 Mar 5. PMID 25740556
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- See also: GLOBOCAN — http://globocan.iarc.fr/Default.aspx
- See also: Population pyramid — https://www.inegi.org.mx/temas/estructura/

DOCUMENTS (1):
  • Informed Consent Form (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT05661292/ICF_000.pdf